CLINICAL TRIAL: NCT04795258
Title: Oral Health Assessment of Children in CP Class in REP/REP+ Areas in the Department of Hérault
Brief Title: Oral Health Assessment of Children in CP Class
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0116
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries
Keywords: Oral hygiene; Public Health; Children; Prevention
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Few oral exams are performed on 6-year-olds (key age for carious disease). This project aims to increase the number of oral check-ups for 6-year-olds in fragile areas (REP/REP+ areas).

ELIGIBILITY:
Inclusion criteria:

* Be a first-grade student enrolled in a school in a zone REP/REP+
* Have a parental permission
* Good understanding of the French language

Exclusion criteria:

- lack of parental permission

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: first-grade student enrolled in a school in a zone REP/REP+
Sampling Method: Non-Probability Sample
Enrollment: 671 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Presence of decay on each tooth present in the mouth | 1 day
  Presence of decay on each tooth present in the mouth
Presence of care on each tooth present in the mouth | 1 day
  Presence of care on each tooth present in the mouth

CONTACTS AND LOCATIONS:
Overall Officials: Camille INQUIMBERT, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC